CLINICAL TRIAL: NCT01254799
Title: Doxycycline in Treatment of Bleeding With DMPA: a Double Blinded Randomized Controlled Trial
Brief Title: Doxycycline in Treatment of Bleeding With Depot Medroxyprogesterone Acetate (DMPA)
Acronym: DOX-DMPA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Omar Mamdouh Shaaban (Other)
Responsible Party: Sponsor-Investigator, Omar Mamdouh Shaaban, Dr, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DOX-DMPA
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-11

CONDITIONS: Uterine Hemorrhage
MeSH Terms: conditions — Uterine Hemorrhage | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Women in this arm will receive identical Placebo capsules twice daily for 5 days
  Interventions: Drug: Placebo
- Doxycycline (Active Comparator): Women in this arm will receive 100 mg doxycycline capsules twice daily for 5 days
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline — 100 mg Doxycycline capsules twice daily for 5 days
  Arms: Doxycycline
Drug: Placebo — Placebo capsules twice daily for 5 days
  Arms: Placebo

SUMMARY:
This study aims to test the effect of Doxycycline in treatment of uterine bleeding during the use of injectable contraception that contains one hormone "progesterone only".

ELIGIBILITY:
Inclusion Criteria:

1. Women under DMPA contraception for at least one month.
2. Accept to participate in the trial after receiving adequate information about the trial including information that she is a part of randomization comprising the possibility of receiving new treatment for bleeding or inactive ingredients.
3. Women's ability to keep an accurate menstrual diary for the study.

Exclusion Criteria:

1. Lactating women for the fear of the effect of tetracycline on the breast-fed infant.
2. Patients with already diagnosed local gynecological abnormality.
3. Women receiving treatment for bleeding within the last one month.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2008-01; Primary Completion 2010-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Stoppage of bleeding within 7 days | 7 days from starting of tretment

SECONDARY OUTCOMES:
Number of days needed to stop a current attack of bleeding | 1 month
Next bleeding free interval | 3 month
Uterine bleeding patterns in the next 3 months after treatment | 3 months
Women satisfaction with the treatment she received | 3 months
Side effects encountered during treatment | 5 days
Discontinuation of the DMPA and its reason | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hany Abdel-Aleem, MD, Principal Investigator — Assiut University; Omar M Shaaban, MD, Study Director — Assiut University; Mahmoud Abdel=Aleem, MD, Study Chair — Assiut University; Gehian N Fetih, PH.D, Study Chair — Faculty of Pharmacy, Assiut University
Locations (1):
- Faculty of Medicine, Asyut, Asyut Governorate, Egypt

REFERENCES:
- [Derived] Abdel-Aleem H, Shaaban OM, Abdel-Aleem MA, Fetih GN. Doxycycline in the treatment of bleeding with DMPA: a double-blinded randomized controlled trial. Contraception. 2012 Sep;86(3):224-30. doi: 10.1016/j.contraception.2012.01.003. Epub 2012 Feb 9. PMID 22325113